CLINICAL TRIAL: NCT07002684
Title: Metabolic Profiling of Esketamine Treatment in Major Depressive Disorder
Brief Title: Metabolic Profiling of Esketamine Treatment in Depressive Disorder
Status: Recruiting | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Tea Fabijanić, MD, Principal Investigator, University of Zagreb
Other Study IDs: 241-25-11-01-1/2-24-2
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients receiving esketamine: patients receiving esketamine
  Interventions: Drug: Esketamine
- healthy controls: no intervention

INTERVENTIONS:
Drug: Esketamine — nasal
  Groups: patients receiving esketamine

SUMMARY:
Major depressive disorder (MDD) is one of the most common psychiatric disorders, characterized by extremely high prevalence, relapse rate and therapeutic resistance. Treatment with ketamine and its enantiomer esketamine is the next step towards the successful treatment and understanding of depression that is resistant to treatment with standard antidepressants. The proposed study will include approximately 50 patients with MDD and 50 healthy control subjects of both sexes. Using untargeted metabolomic approach, we plan to detect changes in biochemical pathways related to the diagnosis of treatment-resistant MDD and changes related to the mechanism of action of esketamine. The proposed research will contribute to further understanding of the mechanism of action of esketamine in patients with MDD. Metabolic changes will be associated with improvements in specific domains of depressive symptoms and symptom severity in subjects with treatment-resistant major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* for healthy control participants: 18-70 years, both sexes, without psychiatric drugs
* for patients: from 18- 70 years, both sexes, failed treatment attempts with at least two antidepressants of the appropriate dose and duration.

Exclusion Criteria:

* for patients: treatment with tryptophan, St. John's wort, and/or opioid analgesics in the last month, daily intake of benzodiazepines;
* for all participants: presence of psychotic symptoms, alcohol and/or drug addiction, disorder seizures, eating disorder, dementia and other neurodegenerative diseases, epilepsy, intellectual disabilities, severe somatic diseases (including insufficiently controlled arterial hypertension, diabetes and thyroid diseases), active psychotherapeutic treatment (except supportive psychotherapy, which is an integral part of every psychiatric treatment and will be the same in all groups of respondents).

Participants will be excluded if they follow a weight loss diet or take weight loss medication, are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical Hospital Centre patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
changed metabolomics | 8 weeks
  Using a non-targeted metabolomic approach, investigate changes in biochemical pathways related to the mechanism of action of the drug esketamine in patients with treatment-resistant major depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Tea Fabijanić, MD, Principal Investigator — University of Zagreb School of Medicine
Locations (1):
- Tea Fabijanić, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No